CLINICAL TRIAL: NCT07061483
Title: Exploring the Impact of Gratitude Journaling for Elementary and Middle School Students
Brief Title: The Impact of Gratitude Journaling in the Classroom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Rhoads (Other)
Responsible Party: Sponsor-Investigator, Michael Rhoads, Assistant Professor of Psychology, Colorado Mesa University
Organization: Colorado Mesa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ColoradoMesa
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Gratitude Journaling; Stress; Belonging; Optimism; Gratitude

STUDY DESIGN:
Intervention Model Description: This study employs a randomized control trial. However, one subgroup of participants were not randomized and only received the treatment condition (gratitude journaling).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (journaling without gratitude) (Placebo Comparator)
  Interventions: Behavioral: Control (journaling without gratitude)
- Experimental (gratitude journaling) (Experimental)
  Interventions: Behavioral: Experimental (Gratitude Journaling)

INTERVENTIONS:
Behavioral: Experimental (Gratitude Journaling) — 60-Day Gratitude Journaling With Guided Prompts
  Arms: Experimental (gratitude journaling)
Behavioral: Control (journaling without gratitude) — 60-Day Journaling Without a Gratitude Focus
  Arms: Control (journaling without gratitude)

SUMMARY:
The objective of this study is to explore the potential benefit of gratitude journaling for students in grades 6-12 and their teachers. Specifically, the investigators seek to determine if the process of gratitude journaling decreases stress, student absenteeism, and teacher burnout, while increasing gratitude, optimism, and a sense of belonging.

DETAILED DESCRIPTION:
Does gratitude journaling decrease perceived stress in students? Does gratitude journaling reduce absenteeism in student class attendance? Does gratitude journaling increase gratitude in participants? Does gratitude journaling increase optimism in participants? Does gratitude journaling increase a sense of belonging in students? And finally, does gratitude journaling decrease teacher burnout? The investigators hypothesize the gratitude journaling process will decrease stress, student absenteeism, and teacher burnout, while increasing gratitude, optimism, and a sense of belonging in participants.

This study will utilize a pre-test post-test correlational study design. As a preliminary pilot study, the investigators seek to determine the potential benefits of gratitude journaling. For this study, Lynnie Gandola is a community partner. The journals were created by Lynnie. The journals she created were supplied to the schools "at cost" with a grant from the School of Life Foundation (schooloflifefoundation.org) as an initiative that principals in the district chose to implement this semester. These journals will be distributed to students regardless of whether or not the pre-test post-test surveys are administered. The investigators are looking to collect data from a journaling exercise that is already taking place. A letter of support from Lynnie Gandola is attached, stating that she approves the assessment of the effectiveness of the gratitude journals. Additionally, this study will use archival class attendance data. This information will be provided as aggregate data from the school districts, with all student information deidentified. For data collection with teachers, a non-randomized control group will also be utilized to compare burnout scores between teacher who did and did not participate in the gratitude journaling.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, individuals must be a student from a school district in the rocky mountain region.

Exclusion Criteria:

* A participant would no longer be eligible for participation if their status as a student ends. Scenarios include incarceration, illegal behavior, or mental illness that requires absence or discontinued school attendance.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 234 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Stress | From enrollment to 60-day post-test
  Perceived Stress Scale. The scale has a range of scores from 0-40 with high scores indicating high stress (low scores are better outcomes).

SECONDARY OUTCOMES:
Gratitude | From enrollment to 60-day post-test
  Gratitude Questionnaire-6. The scale has a range of scores from 6-42 with high scores indicating high gratitude (high scores are better outcomes).
Optimism | From enrollment to 60-day post-test
  Life Orientation Test. The scale has a range of scores from 0-24 with high scores indicating high levels of optimism (high scores are better outcomes).
Belonging | From enrollment to 60-day post-test
  General Belongingness Scale. The scale has a range of scores from 12-84 with high scores indicating high belonging (higher scores are better outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rhoads, PhD, Principal Investigator — Colorado Mesa University
Locations (1):
- Colorado Mesa University, Grand Junction, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The anonymized data set will be uploaded to the OSF data repository.
Time Frame: The IPD is currently available and will be made available as long as OSF manages the data repository.
Access Criteria: The IPD is publicly available.
URL: https://doi.org/10.17605/OSF.IO/JKAXZ

REFERENCES:
- Available data/document: Individual Participant Data Set — https://doi.org/10.17605/OSF.IO/JKAXZ